CLINICAL TRIAL: NCT05647499
Title: Evaluating the Back 2 School Program in a Norwegian Setting: A Multicenter Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tromso (Other)
Collaborators: UiT The Arctic University of Norway (Other); NORCE Norwegian Research Centre AS (Other); Regionsenter for barn og unges psykiske helse (Other); University of Bergen (Other); University of Stavanger (Other); Norwegian University of Science and Technology (Other)
Responsible Party: Principal Investigator, Toril Sorheim Nilsen, Associate Professor, University of Tromso
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UTromso; 779193 (Other: Norsk samfunnsvitenskaplig datatjeneste (NSD))
Record Dates: First submitted 2022-10-30; First posted 2022-12-12 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Absence; School Phobia; Truancy; Socialized; Depression, Anxiety
Keywords: School absence problems; Cognitive behavioral intervention
MeSH Terms: conditions — Phobia, School; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The evaluation of changes in school attendance (primary outcome) following the B2S program will be conducted using a multiple - baseline across subjects' design comparing the individuals' baseline levels of school absenteeism with the level of absenteeism following participation in the B2S program. The structure of the multiple baseline design with 14 subjects is comprised of two treatment conditions, a baseline (control) and an intervention condition with N equally spaced measurement occasions (Hedges, Pustejovsky, & Shadish, 2013). Thus, each subject function as their own control. Changes in secondary outcome measures (psychological wellbeing, school related self-efficacy) are assessed through repeated measurement at pre- (T1), and post intervention (T2).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The Back 2 School program (B2S) for problematic school absenteeism (Experimental): The B2S program is a modular trans-diagnostic cognitive behavioral program aimed at helping children and youth with problematic levels of school absenteeism.
  Interventions: Behavioral: The Back 2 School program for problematic school absenteeism

INTERVENTIONS:
Behavioral: The Back 2 School program for problematic school absenteeism — We will use the Danish version of the revised manual developed within the B2S study in Aarhus, Denmark. The B2S program consists of a 3 to 3,5 -hour initial clinical assessment, a clinical conference, 11 sessions where the youth and/or parent are attending, and a booster session after three months including youth and parent. The B2S manual comprise four school meetings with the child, parents, school staff and therapists present. In the Norwegian pilot study, we will add an extended school module to the B2S-program. The school module includes a pre-meeting interview with the schools in week 1 and session 1 with the school in week 2 or 3. The B2S counselor and the school will decide whether there is a need for an additional meeting between school meetings 1 and 2. There is also a booster session with the child, parents, the school and the B2S team 3 months after the program.
  Other Names: Modular cognitive behavior therapy

SUMMARY:
The goal of this interventional feasibility study is to gain experiences in using the Back 2 School (B2S) program for youth with school attendance problems in Norwegian community school- and health services. The main questions it aims to answer are: • What is the feasibility of the Back 2 School program when implemented in Norwegian community school- and health services? • What are the changes in school attendance rates, measures of psychological difficulties, and school related self-efficacy following the intervention? • How do participants experience the B2S program? 14 youth (10-15 years) with school attendance problems, their caregivers and the school participated in the B2S program provided by an interdisciplinary team during the school term of 2022-2023. Researchers will compare school attendance rates before entrance to the B2S program, at termination of the program and at 3-month follow-up. Also, researchers will compare reports on psychological difficulties, quality of life, and school related-self efficacy at baseline and after the intervention. Researchers investigate participants experiences with the program through qualitative interviews with youths, caregivers, teachers and service providers. The researchers further aim to prepare and establish resources and infrastructure for a large intervention study, and to establish a well-functioning cooperation between researchers, research organizations, and municipalities in different regions.

DETAILED DESCRIPTION:
In Norway, there is no systematic approach for helping youth with school attendance problems. It is important to evaluate potential effective interventions and procedures for these youths. Back 2 School (B2S) is a modular cognitive behavioral intervention for youth with school attendance problems developed and evaluated through a randomized controlled trial by Professor Mikael Thastum and colleagues at the University of Aarhus, Denmark. The theoretical approach of the B2S program is trans-diagnostic, based on a modular cognitive behavior therapy (CBT) manual. The program aims at addressing both school attendance problems and mental health problems that are associated with school absenteeism.

The feasibility study is a collaboration between researchers at the Regional Centers for Child and Youth Mental Health and Child Welfare in Norway (RKBU North, West, Middle and RBUP South/East), and at the University of Bergen, Stavanger, Norwegian University of Science and Technology (NTNU), UiT The Arctic University of Norway, and the University of Aarhus, Denmark.

In a nationwide feasibility study in Norway, B2S is evaluated in 8 municipalities during the school term of 2022-2023. Participants was 14 young people (10-15 years), their parents/caregivers and their school.

The feasibility study has several aims. One overall aim is to gain experience in using the Back 2 School program in Norwegian community school- and health services and to assess the the feasibility of the program in those settings. Another aim is to prepare and establish resources and infrastructure for a larger intervention study, and to establish a well-functioning cooperation between researchers, research organizations, and municipalities in different regions. Also, questions regarding the process of implementation of the program in community service settings will be an important issue for the study.

By using a mixed method approach the study will combine quantitative and qualitative methods addressing the following research questions:

Quantitative:

1. What are the characteristics of youths with SA and their families?
2. What are the changes in school absence rate, school related self-efficacy, and psychological difficulties following the intervention?
3. What additional needs for interventions and services are identified at termination of the program?
4. What is the degree of drop out, and level of satisfaction with the B2S program among children, parents and teachers?

   Qualitative:
5. How do children, youths and their caregivers experience the B2S program? In what ways has the intervention been helpful? Are there ways the program and service system should be changed to better fit the needs of the youth and families struggling with SA? What would be optimized treatment and services for this group?
6. How do the team of professionals experience working with the B2S program to help children and youth with problematic SA? How did the professionals experience the training, the manual and the supervision? Are there ways the program and service system should be changed to better fit the needs of the youngster and families struggling with SA? What do the therapists consider to be optimized treatment and services for this group?
7. How do school staff experience the B2S program and the extended school module?

Based on the findings from the pilot study the aim is to answer the following questions:

* How should a larger-scale implementations study of the Back 2 School program be planned, optimized and conducted?
* What should be the treatment comparison condition?
* What is an optimal level of school involvement in B2S?

Project period Data for the feasibility study was collected during the school year of 2022 -2023. The analysis of the results and writing of reports are under actual preparation in 2024. The project group are currently applying for funding of the national effectiveness and implementation study, the main study.

The 5- day training of the professionals in the B2S program took place in March 2022. Beforehand, the teams have recruited a case for the first implementation of the program (the rehearsal case). The data collected during the rehearsal case is not included in the database of the pilot. From September/October 2022 through June 2023 each team will conduct the B2S program and collect data from two cases each.

Methods:

Participants and settings:

14 youth (10-15 years of age) was included in the feasibility study. The study was conducted in eight Norwegian municipalities. Each region (East, West, Middle, North) recruited one to two teams of professionals from their geographical area. The setting for the B2S intervention was within first line services in the municipalities that are imposed to provide services for the target group.

Procedure:

Therapists Each municipality formed a B2S Team consisting of three professionals. The teams were interdisciplinary including both member(s) with a relevant health profession (clinical psychologist, medical doctor, health nurse, social educator) and member(s) within a pedagogical profession (teacher, special educator).

Training All professionals received a 5-days training course comprising assessment measures and proceedings, case formulation and the Back 2 School manual. Following training, the teams had weekly supervision by an interdisciplinary team of supervisors, consisting of 1 CBT expert and one with educational professional background, to ensure adherence and quality in delivery. Professionals providing the B2S intervention received a total of 70 hours of training (35 hours) and supervision (estimated 35 hours) during the pilot study.

Recruitment Children and youth with problematic school absenteeism (defined as above 10% absence during the last 3 months of school) that were referred to communal services was invited to a information meeting regarding the B2S intervention. Children and/or caregivers that for whatever reason was not eligible for the B2S program were assigned the communal service´s ordinary measures. Children and caregivers that met inclusion criteria and did not meet exclusion criteria, and that wished to sign up for the intervention, were included in the feasibility study.

Assessment All data collection and assessment within the pilot study were obtained for two main aims: 1) To inform intervention planning and adjustment of the intervention when implementing the B2S program with each individual youth and family, and 2) To answer the research questions of the pilot study.

All assessments within the pilot study were collected on paper forms. Children, parents/caregivers and teachers filled out separate forms. At inclusion to the pilot study, the youth, parents and teachers immediately started to register school absence (primary outcome) daily on paper form. The Back 2 School team sent the T1 collection of questionnaires on paper forms to the families by post or the questionnaires were handed to the families when they signed the informed consent to participate in the pilot study. Youth aged ≤ 11 years could fill out the questionnaire themselves. Children aged 8 to 10 years filled out the questionnaire with the aid from the B2S counselor/team.

Clinical interview and case formulation The intervention starts with the families attending a 3-3.5-hour clinical interview that consists of a range of structured questions. The interview aims to achieve an understanding of the youngster's school absenteeism, development, the family and social situation, and functioning in daily life. The interview also includes a structured joint youth and parent interview developed for the B2S program to assess type and degree of potential mental health problems in the youth.

Following the initial assessment, a case-formulation according is developed in cooperation between the B2S counselor/team and the family. The case formulation is based on the qualitative and quantitative information from the interviews and the baseline measures.

The family and B2S counselor/team identify the motivational function of the child's school absenteeism, which decides which module in the program that will best fit the individual youth and his/her family. When school absenteeism is identified as motivated by positive reinforcement for not attending, CBT procedures targeting parent management and contingency management to minimize the incentives for absenteeism and augment incentives for attendance are indicated. School absenteeism identified as motivated by negative reinforcement for attending school involves CBT procedures such as cognitive restructuring, and exposure-based interventions to reduce anxious or depressive symptoms. The manual includes and targets both specific school attendance problems related tasks, and symptom-specific modules targeting sub-clinical or clinical levels of anxiety, depression, or behavioral problems. During the first two weeks of the intervention, there are two weekly sessions to emphasize the importance of immediately increasing school attendance. The following 6 sessions include weekly or biweekly sessions as appropriate for each family. The conducting of the booster session is flexible regarding the timing and will be held within 3 months after the last session.

The school module: Collaborating with the school is important in the B2S and four meetings with teachers from the youth's school, the therapist, and parents and also a booster session 3 months after the program are included in the manual. In the feasibility study, an extended school module developed for this study was implemented to include the schools from the beginning of the program to facilitate a positive school environment for the child and collaboration between the school and the family. The school module includes a pre-meeting interview with the schools in week 1 and session 1 with the school in week 2 or 3. These are in addition to the sessions described in the Danish manual. The B2S counselor/team and the school will decide whether there is a need for an additional meeting between school meetings 1 and 2 and.

ELIGIBILITY:
Inclusion Criteria:

1. Youth enrolled in a public school within the municipality,
2. aged 6-16 years and in 1st to -10th grade (excluding second semester of the 10th grade),
3. having a level of school absenteeism above 10% during the last 3 months of school (excluding legal absence, e.g., permitted extra holidays),
4. The youth and at least one parent/caregiver understand and speak Norwegian sufficiently to participate in the intervention and complete questionnaires,
5. At minimum one of the parents is motivated for working on increasing the youth's school attendance,
6. The participating families are willing to record baseline levels of school absenteeism and to participate in assessment, intervention procedures, and follow-up assessment,
7. Written informed consent from caregiver with judicial parental rights and responsibilities (usually both parents) to take part in the B2S pilot study is obtained.

Exclusion Criteria:

* Youth with a diagnosis of autism spectrum disorders cannot be included in the pilot study (exclusion criteria). Also, youth in need of acute and/or more intensive specialist mental health services (e.g., due to suicidal risk, ongoing symptoms of psychosis, ongoing eating disorder) cannot be included.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Change in School absence data | 2 weeks prior to initiation of the program (T1), 2 weeks prior to the finalization of the program (T2) and 2 weeks prior to the 3-month follow-up meetings (T3).
  The primary outcome measure is change in school absence data registered on paper-form on a daily basis by teachers, parents' and youths. The informants register presence/absence session by session during their school day, including a remark on presence according to their individual schedule. Official school record absence data is recorded retrospectively during a period of 2 weeks prior to initiation of the program (T1), 2 weeks prior to the finalization of the program (T2) and 2 weeks prior to the 3-month follow-up meetings (T3).

SECONDARY OUTCOMES:
The Strengths and Difficulties Questionnaire (SDQ-C/P/T) | At baseline, and up to 12 weeks (at termination)
  The SDQ (Goodman, 1997) is a 25- item screening instrument covering emotional, behavioral and social difficulties, peer relations, prosocial behavior, as well as five questions regarding functional impairment in children and adolescents (2 - 17 years of age). Both the self-report version (from age 11), and the parent- and teacher- report versions will be used. A total problem score,five problem sub-scales and a prosocial behavior scale are computed. Higher scores indicate higher levels of problem on the problem scales, and higher level of prosocial behavior on the prosocial behavior sub-scale
The Spence Children's Anxiety Scale (SCAS C/P) | At baseline, and at up to 12 weeks (at termination)
  The SCAS (Spence, 1998) is a self-report and parent reported rating scale with 38 items (child version includes additional six positive filler items) regarding symptoms of anxiety rated on a 4-point scale. SCAS consists of six sub-scales: social phobia (six items), panic disorder and agoraphobia (nine items), generalized anxiety disorder (six items), obsessive-compulsive disorder (six items), separation anxiety disorder (six items), and fear of physical injury /simple phobia (five items). Both the youth (SCAS-C) and the parent version (SCAS-P) will be used. Raw scores are converted into T-scores with an average of 50 and SD of 10. Higher scores indicate higher levels of anxiety symptoms.
The Mood and Feelings Questionnaire (MFQ C/P) | At baseline, and up to 12 weeks (at termination)
  The MFQ (Angold et al., 1995; Costello & Angold, 1988) is a 33-item screening tool for depression in youths aged 6 to 19 years. In the pilot study we use the short version of the MFQ with 13 items. The MFQ includes a youth (MFQ-C) and a parent version (MFQ-P). Scores are summed and high scores indicated higher levels of depressive symptoms.
The Self-efficacy Questionnaire for School Situations (SEQ-SS) | At baseline, and up to 12 weeks (at termination)
  SEQ-SS (Heyne, 1998) was developed to assess the expectations of school-refusing youth concerning self-efficacy. The SEQ-SS consists of 12 items, and 2 sub-scales: Academic/Social Stress and Separation/Discipline Stress.A total score is derived by summing the different items, yielding scores from 12-60 points, with higher scores reflecting greater self-efficacy.
The Self-efficacy Questionnaire Responding to School Attendance Problems (SEQ-RSAP) | At baseline, and up to 12 weeks (at termination)
  SEQ-RSAP (Heyne, Maric, & Westenberg, 2007) was developed to assess parents' self-efficacy regarding helping their child to attend school regularly and without difficulty. A total score is derived by summing the 25 items, yielding scores between 25 and 100. Higher scores reflect higher self efficacy for responding to SAP.
About being bullied | At baseline, and up to 12 weeks (at termination)
  Bullying (Olweus, 1993) register the youths' personal experience of being bullied through 2 items. Bullying will be defined as "a student is being bullied when he or she is exposed repeatedly over time to negative and hurtful actions on the part of one or more students. It is difficult for the student being bullied to defend himself or herself. Bullying may take place frequently or infrequently. Bullying can be verbal (e.g., name-calling, threats), physical (e.g., hitting) or psychological (e.g., rumors, shunning/exclusion). It is bullying when someone is teasing repeatedly in a mean or hurtful way" (Olweus, 1993).
The Family Assessment Device (FAD) | At baseline, and up to 12 weeks (at termination)
  FAD (Epstein, Baldwin, & Bishop, 1983) was developed to assess dimensions of family function. It consists of three sub-scales, with 60 statements describing various aspects of family functioning. FAD is designed to be completed by family members over the age of 12 years. Scoring is on a 4-point scale (from 1 for strongly agree to 4 for strongly disagree) with the scale for the negatively worded items reversed. Scoring is on a 4-point scale (from 1 for strongly agree to 4 for strongly disagree) with the scale for the negatively worded items reversed. The total score is then divided by the number of items on the sub-scale giving a total score ranging from 1.0 (best functioning) to 4.0 (worse functioning).
KIDSCREEN-27 | At baseline, and up to 12 weeks (at termination)
  KIDSCREEN-27 (Ravens-Sieberer, 2006) is a 27-item scale used to assess generic health-related quality of life. The KIDSCREEN comes in a child version and a parent proxy-version. The scale has five dimensions: Physical Well-Being, Psychological Well-Being, Autonomy & Parents, Peers & Social Support and School Environment. Raw Scores are converted in to T-scores with an average of 50 and SD 10. Higher scores reflect higher levels of QoL.

CONTACTS AND LOCATIONS:
Overall Officials: Frode Adolfsen, PHD, Study Chair — UiT; Kristin G Askeland, PHD, Study Chair — NORCE Norwegian Research Centre AS; Simon P Neumer, PHD, Study Chair — Regionssenter for barn og unge
Locations (4):
- Norway (4):
  - NORCE research center, Bergen
  - Regionssenter for barn og unge (RBUP), Oslo
  - UiT The Arctic University Norway, Tromsø
  - Norges Tekniske Naturvitenskapelige Universitet, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Epstein, N. B., Baldwin, L. M., & Bishop, D. S. (1983). The McMaster Famility Assessment Device. Journal of Marital and Family Therapy, 9(2), 171-180.
- [Background] Heyne, D., Maric, M., & Westenberg, M. (2007). "Self-Efficacy Questionnaire for Responding to School Attendance Problems" Unpublished measure. Leiden the Netherlands.
- [Background] Ravens-Sieberer U. [Special aspects of the quality of life of children]. Dtsch Med Wochenschr. 2006 May 12;131(19 Suppl 1):S27-30. doi: 10.1055/s-2006-941737. German. PMID 16688662
- [Background] Thastum M, Johnsen DB, Silverman WK, Jeppesen P, Heyne DA, Lomholt JJ. The Back2School modular cognitive behavioral intervention for youths with problematic school absenteeism: study protocol for a randomized controlled trial. Trials. 2019 Jan 8;20(1):29. doi: 10.1186/s13063-018-3124-3. PMID 30621787
- [Result] Goodman R. The Strengths and Difficulties Questionnaire: a research note. J Child Psychol Psychiatry. 1997 Jul;38(5):581-6. doi: 10.1111/j.1469-7610.1997.tb01545.x. PMID 9255702
- [Result] Costello EJ, Angold A. Scales to assess child and adolescent depression: checklists, screens, and nets. J Am Acad Child Adolesc Psychiatry. 1988 Nov;27(6):726-37. doi: 10.1097/00004583-198811000-00011. No abstract available. PMID 3058677
- [Result] Spence SH. A measure of anxiety symptoms among children. Behav Res Ther. 1998 May;36(5):545-66. doi: 10.1016/s0005-7967(98)00034-5. PMID 9648330
- [Result] Heyne, D., King, N., Tonge, B., Rollings, S., Pritchard, M., Young, D., & Myerson, N. (1998). The self-efficacy questionnaire for school situations: Development and psychometric evaluation. Behaviour Change, 15(1), 31-40. https://doi.org/10.1017/S081348390000588X
- [Result] Jeppesen P, Wolf RT, Nielsen SM, Christensen R, Plessen KJ, Bilenberg N, Thomsen PH, Thastum M, Neumer SP, Puggaard LB, Agner Pedersen MM, Pagsberg AK, Silverman WK, Correll CU. Effectiveness of Transdiagnostic Cognitive-Behavioral Psychotherapy Compared With Management as Usual for Youth With Common Mental Health Problems: A Randomized Clinical Trial. JAMA Psychiatry. 2021 Mar 1;78(3):250-260. doi: 10.1001/jamapsychiatry.2020.4045. PMID 33355633

DOCUMENTS (1):
  • Study Protocol (2022-10-21): https://cdn.clinicaltrials.gov/large-docs/99/NCT05647499/Prot_000.pdf